CLINICAL TRIAL: NCT06990451
Title: Effect of Time Pressure Motor Training With Step Square Exercise on Decision Making Ability and Quality of Life in Stroke Patients
Brief Title: Time Pressure Motor Training With Step Square Exercise on Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Lama Saad El-Din Mahmoud, Assistant Professor of Neurology and Neurosurgery Faculty of Physical Therapy October 6 University, October 6 University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005777
Record Dates: First submitted 2025-05-18; First posted 2025-05-25 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Time Pressure motor management with step square exercise
  Interventions: Other: time pressure; Other: step square exercise; Other: functional care training
- control group (Experimental): conventional treatment
  Interventions: Other: functional care training

INTERVENTIONS:
Other: time pressure — a set of alternative cognitive strategies that allow patients in real-life tasks to compensate for their mental slowness
  Arms: study group
Other: step square exercise — is a form of highly specific balance training for falls prevention which directly addresses stepping capacity-a commonly executed protective strategy for maintaining balance in the everyday environment
  Arms: study group
Other: functional care training — Intensive functional endurance, strength, and balance exercises, and selected physical therapy interventions for balance

SUMMARY:
to investigate The Efficacy of Time Pressure motor rehabilitation with step square exercise (SEE) on decision making ability & quality of life in stroke Patients

DETAILED DESCRIPTION:
PURPOSE: to investigate The Efficacy of Time Pressure motor rehabilitation with step square exercise (SEE) on decision making ability & quality of life in stroke Patients BACKGROUND: stroke patients demonstrate impairments in decision making ability leads to deficits in patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

* age from 50 to 65 years old
* both Sex
* the duration of illness more than three months
* post stroke hemiplegia
* mild spasticity ranged from (1:1+) according to Modified Ashworth Scale

Exclusion Criteria:

* stroke occurred less than 3 months ago
* Patients with severe cognitive or psychiatric impairment aphasia who could not understand the instructions given to him by physical therapist or unable to perform the task
* any other orthopedic disorders or neurologic diseases.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
The Trail Making Test | four weeks
  he Trail Making Test for assessing decision making ability
Mini-Mental State Exam | four weeks
  Mini-Mental State Exam: that tests five areas of cognitive function: orientation, registration, attention and calculation, recall, and language.

SECONDARY OUTCOMES:
Stroke Specific Quality of Life | four weeks
  The Stroke Specific Quality Of Life scale (SS-QOL) is a patient-centered outcome measure intended to provide an assessment of health-related quality of life (HRQOL) specific to patients with stroke.
The Functional Independence Measure | four weeks
  The Functional Independence Measure (FIM) is an instrument that was developed as a measure of disability for a variety of populations and is not specific to any diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Lama Saad El-Din Mahmoud, Al Jīzah, Select State, Egypt